CLINICAL TRIAL: NCT04559880
Title: Tranexamic Acid to Prevent Bleeding After Endoscopic Resection of Large Colorectal Polyps: A Pilot Project
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lawrence Charles Hookey (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor-Investigator, Lawrence Charles Hookey, Director, Endoscopy, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6029804
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Polyp, Colorectal
Keywords: Endoscopic Mucosal Resection (EMR); Tranexamic Acid; Colonoscopy
MeSH Terms: conditions — Polyps | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: 25 consecutive patients treated with tranexamic acid after endoscopic mucosal resection (EMR) of large non-pedunculated colorectal polyps (LNPCP's) to prevent post-polypectomy delayed bleeding (PPDB).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tranexamic Acid (Experimental): Intra-procedural tranexamic acid (TXA) - 1 gram, IV
  Post-procedural tranexamic acid (TXA) - 1 gram, oral, three times per day for 5 days
  Interventions: Drug: Tranexamic Acid Injection [Cyklokapron]

INTERVENTIONS:
Drug: Tranexamic Acid Injection [Cyklokapron] — Intra-procedurally, participants will receive 1 gram of intravenous tranexamic acid immediately following the polypectomy. Participants will also take oral tranexamic acid tablets (three times per day) at home for the five days following the procedure.
  Other Names: Tranexamic Acid Oral Tablets [Cyklokapron]

SUMMARY:
Colorectal cancer is the second most common cancer in Canada. Colonoscopy and removal of precancerous polyps (polypectomy) reduces the incidence and mortality associated with colorectal cancer. However, polypectomy is associated with adverse events. Post-polypectomy bleeding has a significant impact on the life of the patient as it can require hospitalization, transfusions, repeat colonoscopy and rarely death. It is also a substantial cost to the health care system. There currently is no standard of care to prevent bleeding after polypectomy.

Tranexamic acid reduces fibrinolysis by slowing down the conversion of plasminogen to plasmin which may prevent bleeding. Although this medication is used extensively for other purposes, it has not been studied before to prevent post-polypectomy bleeding.

This pilot study will examine factors involved in the feasibility of conducting a large-scale randomized controlled trial (RCT). This pilot study will include 25 consecutive patients who are treated with tranexamic acid after endoscopic mucosal resection (EMR) of large non-pedunculated colorectal polyps (LNPCP's) to prevent PPDB.

DETAILED DESCRIPTION:
Colorectal cancer is the second most common cancer in Canada. Colonoscopy and removal of precancerous polyps (polypectomy) reduces the incidence and mortality associated with colorectal cancer. However, polypectomy is associated with adverse events. Post-polypectomy bleeding has a significant impact on the life of the patient as it can require hospitalization, transfusions, repeat colonoscopy and rarely death. It is also a substantial cost to the health care system. Post-polypectomy delayed bleeding (PPDB) can occur up to a month following the procedure but is typically seen within the first week. Risk factors include the size of the polyp, antithrombotic or anticoagulation use, age, major comorbidities and proximal colon polyps. The incidence of bleeding after removal of large polyps is estimated to be around 2.6%-9.7%. There currently is no standard of care to prevent bleeding after polypectomy. Tranexamic acid reduces fibrinolysis by slowing down the conversion of plasminogen to plasmin which may prevent bleeding.

This pilot study will examine factors involved in the feasibility of conducting a large-scale RCT. This pilot study will include 25 consecutive patients who are treated with tranexamic acid after endoscopic mucosal resection (EMR) of large non-pedunculated colorectal polyps (LNPCP's) to prevent PPDB.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 who have non-pedunculated colorectal polyps,
2. Polyps ≥2cm,
3. Polyps removed by endoscopic mucosal resection (EMR),
4. Agree to be followed up by phone,
5. Ability to read and understand the English language.

Exclusion Criteria:

1. Patients who have inflammatory bowel disease,
2. Diagnosed bleeding disorder,
3. Ulcerated morphology of polyps or those with proven invasive cancer,
4. Patients with a history of or are at higher risk of thromboembolic events (atrial fibrillation on anticoagulation, history of stroke, transient ischemic attack (TIA), pulmonary embolism, deep vein thrombosis, hypercoagulable state, oral contraceptive pill (OCP) or hormone replacement therapy use, mechanical heart valve on anticoagulation, myocardial infarction in the last twelve months, retinal vein or retinal artery occlusion),
5. Unable to provide follow up,
6. Unable to provide consent,
7. Pregnancy,
8. Patients undergoing endoscopic submucosal dissection (ESD),
9. Seizure disorder,
10. Ureteral obstruction within past 6 months,
11. Subarachnoid hemorrhage within past 6 months,
12. A diagnosed acquired defective colour vision disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Enrollment frequency | Through study completion, an average of 6 months
  How many participants are enrolled each week
Study drug compliance rates | Through study completion, an average of 6 months
  Number of participants that receive the intravenous tranexamic acid within 2 hours of polyp removal and the number of participants that receive every scheduled dose of the tranexamic acid at home
Recruitment rates | Through study completion, an average of 6 months
  How many eligible patients decide to participate in the study
Follow-up rates | Through study completion, an average of 6 months
  How many participants complete all follow-up phone calls

SECONDARY OUTCOMES:
Adverse events | Up to 30 days
  How many participants experience thromboembolic events, perforation and post-polypectomy electrocoagulation syndrome, seizure activity and vision changes
Post-procedure bleeding | Up to 30 days
  How many participants experience severe bleeding event that requires hospitalization, transfusion, colonoscopy, surgery or another invasive intervention within 30 days after completion of the colonoscopy with polypectomy

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bechara, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre - Hotel Dieu Hospital Site, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nishihara R, Wu K, Lochhead P, Morikawa T, Liao X, Qian ZR, Inamura K, Kim SA, Kuchiba A, Yamauchi M, Imamura Y, Willett WC, Rosner BA, Fuchs CS, Giovannucci E, Ogino S, Chan AT. Long-term colorectal-cancer incidence and mortality after lower endoscopy. N Engl J Med. 2013 Sep 19;369(12):1095-105. doi: 10.1056/NEJMoa1301969. PMID 24047059
- [Result] ASGE Standards of Practice Committee; Fisher DA, Maple JT, Ben-Menachem T, Cash BD, Decker GA, Early DS, Evans JA, Fanelli RD, Fukami N, Hwang JH, Jain R, Jue TL, Khan KM, Malpas PM, Sharaf RN, Shergill AK, Dominitz JA. Complications of colonoscopy. Gastrointest Endosc. 2011 Oct;74(4):745-52. doi: 10.1016/j.gie.2011.07.025. No abstract available. PMID 21951473
- [Result] Albeniz E, Fraile M, Ibanez B, Alonso-Aguirre P, Martinez-Ares D, Soto S, Gargallo CJ, Ramos Zabala F, Alvarez MA, Rodriguez-Sanchez J, Mugica F, Nogales O, Herreros de Tejada A, Redondo E, Pin N, Leon-Brito H, Pardeiro R, Lopez-Roses L, Rodriguez-Tellez M, Jimenez A, Martinez-Alcala F, Garcia O, de la Pena J, Ono A, Alberca de Las Parras F, Pellise M, Rivero L, Saperas E, Perez-Roldan F, Pueyo Royo A, Eguaras Ros J, Zuniga Ripa A, Concepcion-Martin M, Huelin-Alvarez P, Colan-Hernandez J, Cubiella J, Remedios D, Bessa I Caserras X, Lopez-Viedma B, Cobian J, Gonzalez-Haba M, Santiago J, Martinez-Cara JG, Valdivielso E, Guarner-Argente C; Endoscopic Mucosal Resection Endoscopic Spanish Society Group. A Scoring System to Determine Risk of Delayed Bleeding After Endoscopic Mucosal Resection of Large Colorectal Lesions. Clin Gastroenterol Hepatol. 2016 Aug;14(8):1140-7. doi: 10.1016/j.cgh.2016.03.021. Epub 2016 Mar 24. PMID 27033428
- [Result] Pohl H, Grimm IS, Moyer MT, Hasan MK, Pleskow D, Elmunzer BJ, Khashab MA, Sanaei O, Al-Kawas FH, Gordon SR, Mathew A, Levenick JM, Aslanian HR, Antaki F, von Renteln D, Crockett SD, Rastogi A, Gill JA, Law RJ, Elias PA, Pellise M, Wallace MB, Mackenzie TA, Rex DK. Clip Closure Prevents Bleeding After Endoscopic Resection of Large Colon Polyps in a Randomized Trial. Gastroenterology. 2019 Oct;157(4):977-984.e3. doi: 10.1053/j.gastro.2019.03.019. Epub 2019 Mar 15. PMID 30885778
- [Result] Feagins LA. Colonoscopy, Polypectomy, and the Risk of Bleeding. Med Clin North Am. 2019 Jan;103(1):125-135. doi: 10.1016/j.mcna.2018.08.003. Epub 2018 Nov 1. PMID 30466669
- [Result] Hassan C, Repici A, Sharma P, Correale L, Zullo A, Bretthauer M, Senore C, Spada C, Bellisario C, Bhandari P, Rex DK. Efficacy and safety of endoscopic resection of large colorectal polyps: a systematic review and meta-analysis. Gut. 2016 May;65(5):806-20. doi: 10.1136/gutjnl-2014-308481. Epub 2015 Feb 13. PMID 25681402
- [Result] Burgess NG, Metz AJ, Williams SJ, Singh R, Tam W, Hourigan LF, Zanati SA, Brown GJ, Sonson R, Bourke MJ. Risk factors for intraprocedural and clinically significant delayed bleeding after wide-field endoscopic mucosal resection of large colonic lesions. Clin Gastroenterol Hepatol. 2014 Apr;12(4):651-61.e1-3. doi: 10.1016/j.cgh.2013.09.049. Epub 2013 Oct 1. PMID 24090728
- [Result] Forbes N, Frehlich L, James MT, Hilsden RJ, Kaplan GG, Wilson TA, Lorenzetti DL, Tate DJ, Bourke MJ, Heitman SJ. Routine Prophylactic Endoscopic Clipping Is Not Efficacious in the Prevention of Delayed Post-Polypectomy Bleeding: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Can Assoc Gastroenterol. 2019 Aug;2(3):105-117. doi: 10.1093/jcag/gwy033. Epub 2018 Jul 20. PMID 31294373
- [Result] Albeniz E, Alvarez MA, Espinos JC, Nogales O, Guarner C, Alonso P, Rodriguez-Tellez M, Herreros de Tejada A, Santiago J, Bustamante-Balen M, Rodriguez Sanchez J, Ramos-Zabala F, Valdivielso E, Martinez-Alcala F, Fraile M, Elosua A, Guerra Veloz MF, Ibanez Beroiz B, Capdevila F, Enguita-German M. Clip Closure After Resection of Large Colorectal Lesions With Substantial Risk of Bleeding. Gastroenterology. 2019 Nov;157(5):1213-1221.e4. doi: 10.1053/j.gastro.2019.07.037. Epub 2019 Jul 27. PMID 31362007
- [Result] Roberts I, Shakur H, Coats T, Hunt B, Balogun E, Barnetson L, Cook L, Kawahara T, Perel P, Prieto-Merino D, Ramos M, Cairns J, Guerriero C. The CRASH-2 trial: a randomised controlled trial and economic evaluation of the effects of tranexamic acid on death, vascular occlusive events and transfusion requirement in bleeding trauma patients. Health Technol Assess. 2013 Mar;17(10):1-79. doi: 10.3310/hta17100. PMID 23477634
- [Result] WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 27;389(10084):2105-2116. doi: 10.1016/S0140-6736(17)30638-4. Epub 2017 Apr 26. PMID 28456509
- [Result] Bennett C, Klingenberg SL, Langholz E, Gluud LL. Tranexamic acid for upper gastrointestinal bleeding. Cochrane Database Syst Rev. 2014 Nov 21;2014(11):CD006640. doi: 10.1002/14651858.CD006640.pub3. PMID 25414987
- [Result] Smith SR, Murray D, Pockney PG, Bendinelli C, Draganic BD, Carroll R. Tranexamic Acid for Lower GI Hemorrhage: A Randomized Placebo-Controlled Clinical Trial. Dis Colon Rectum. 2018 Jan;61(1):99-106. doi: 10.1097/DCR.0000000000000943. PMID 29215478
- [Result] Grass F, Braafladt S, Alabbad J, Lovely JK, Kelley SR, Mathis KL, Huebner M, Larson DW. The effects of tranexamic acid on blood loss and transfusion rate in colorectal surgery. Am J Surg. 2019 Nov;218(5):876-880. doi: 10.1016/j.amjsurg.2019.03.013. Epub 2019 Mar 15. PMID 30926155